CLINICAL TRIAL: NCT05556265
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 2 Study to Evaluate Clinical Efficacy and Safety of Deucravacitinib (BMS-986165) in Participants With Alopecia Areata
Brief Title: A Study to Evaluate Efficacy and Safety of Deucravacitinib in Participants With Alopecia Areata
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM011-134; U1111-1246-1767 (Registry Identifier: WHO); 2020-000113-33 (EudraCT Number)
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Alopecia Areata
Keywords: Deucravacitinib; IM011134; BMS-986165
MeSH Terms: conditions — Alopecia Areata | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Deucravacitinib Dose 1 (Experimental)
  Interventions: Drug: Deucravacitinib; Other: Placebo
- Deucravacitinib Dose 2 (Experimental)
  Interventions: Drug: Deucravacitinib; Other: Placebo
- Placebo, followed by Deucravacitinib Dose 1 or Dose 2. (Placebo Comparator)
  Interventions: Drug: Deucravacitinib; Other: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Other Names: BMS-986165
Other: Placebo — Placebo was administered.

SUMMARY:
The purpose of this study is to evaluate the efficacy of deucravacitinib versus placebo at Week 24 and safety and tolerability of deucravacitinib versus placebo in adults with alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis of alopecia areata (AA) for at least 6 months.
* Current episode of scalp hair loss (at screening) must meet the following criteria: duration at least 6 months; duration of current hair loss episode of AA affecting ≥ 50% of the scalp not exceeding 8 years; scalp hair loss has been stable (no significant spontaneous regrowth [> 10%] over the last 6 months)
* SALT score ≥ 50 at Screening and Day 1. Participant with complete scalp hair loss (SALT score of 100) with or without body hair involvement can be included.

Exclusion Criteria:

* Participant with diffuse-type AA or other forms of hair loss, including traction alopecia, lichen planopilaris, central centrifugal cicatricial alopecia, frontal fibrosing alopecia, etc.
* Other active skin diseases affecting the scalp that in the opinion of the investigator may interfere with accurate assessment of SALT score.
* Extensive tattooing of the scalp that, in the opinion of the investigator, may interfere with the accurate assessment of SALT score.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (28):
- United States (12):
  - Local Institution - 0016, Santa Monica, California
  - Local Institution - 0036, New Haven, Connecticut
  - Local Institution - 0018, Tampa, Florida
  - Local Institution - 0023, Clinton Township, Michigan
  - Local Institution - 0024, New York, New York
  - Local Institution - 0019, Chapel Hill, North Carolina
  - Local Institution - 0011, Portland, Oregon
  - Local Institution - 0032, Pittsburgh, Pennsylvania
  - Local Institution - 0012, Austin, Texas
  - Local Institution - 0013, Houston, Texas
  - Local Institution - 0014, San Antonio, Texas
  - Local Institution - 0017, South Jordan, Utah
- Australia (2):
  - Local Institution - 0003, Kogarah, New South Wales
  - Local Institution - 0005, Carlton, Victoria
- Canada (6):
  - Local Institution - 0015, Winnipeg, Manitoba
  - Local Institution - 0021, Markham, Ontario
  - Local Institution - 0009, Peterborough, Ontario
  - Local Institution - 0010, Richmond Hill, Ontario
  - Local Institution - 0034, Montreal, Quebec
  - Local Institution - 0027, Québec, Quebec
- France (2):
  - Local Institution - 0033, Nice
  - Local Institution - 0020, Paris
- Japan (4):
  - Local Institution - 0031, Hamamatsu
  - Local Institution - 0028, Kōtoku
  - Local Institution - 0030, Mitaka-Shi
  - Local Institution - 0029, Shinjuku-Ku
- Poland (2):
  - Local Institution - 0026, Wroclaw, Lower Silesian Voivodeship
  - Local Institution - 0025, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated due to change in business objectives.
Pre-assignment Details: 94 participants randomized and treated in Placebo controlled period. the 31 participants in the placebo cohort, were re-randomized into the active treatment cohort.
Groups:
- Deucravacitinib 6 mg QD: Participants with alopecia areata received deucravacitinib 6 mg tablet orally once daily (QD) from Day 1 to Week 24 in Placebo-controlled Period.
- Deucravacitinib 6 mg BID: Participants with alopecia areata received deucravacitinib 6 mg tablet orally twice daily (BID) from Day 1 to Week 24 in Placebo-controlled Period.
- Placebo: Participants with alopecia areata received placebo tablet orally twice daily (BID) from Day 1 to Week 24 in Placebo-controlled Period.
- Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD: Participants initially randomized to receive placebo in Placebo-controlled Period were re-randomized to this arm at the Week 24 visit. Participants in this arm received 6 mg deucravacitinib tablet orally QD till Week 52 in Active Treatment Period.
- Active-Treatment Period: Placebo Followed by Deucravacitinib 6 mg BID: Participants initially randomized to receive placebo in Placebo-controlled Period were re-randomized to this arm at the Week 24 visit. Participants in this arm received 6 mg deucravacitinib tablet orally BID till Week 52 in Active Treatment Period.
Period: Placebo-Controlled (Day 1 to Week 24)
Arm/Group | Deucravacitinib 6 mg QD | Deucravacitinib 6 mg BID | Placebo | Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD | Active-Treatment Period: Placebo Followed by Deucravacitinib 6 mg BID
Started | 32 | 31 | 31 | 0 | 0
Completed | 32 | 26 | 31 | 0 | 0
Not Completed | 0 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Participant request to discontinue study treatment | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 0
Period: Active Treatment (Week 25 to Week 52)
Arm/Group | Deucravacitinib 6 mg QD | Deucravacitinib 6 mg BID | Placebo | Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD | Active-Treatment Period: Placebo Followed by Deucravacitinib 6 mg BID
Started | 32 | 26 | 0 | 16 (16 out of 31 participants from Placebo arm (Placebo-controlled Period) re-randomized to this arm in Active Treatment period.) | 15 (15 out of 31 participants from Placebo arm (Placebo-controlled Period) re-randomized to this arm in Active Treatment Period.)
Completed | 8 | 5 | 0 | 5 | 3
Not Completed | 24 | 21 | 0 | 11 | 12
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 3 | 1
Not completed — Participant request to discontinue study treatment | 1 | 3 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 19 | 12 | 0 | 6 | 9
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deucravacitinib 6 mg QD | Deucravacitinib 6 mg BID | Placebo | Total
Number analyzed (Participants) | 32 | 31 | 31 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (13.37) | 43.4 (13.81) | 38.9 (14.40) | 39.4 (14.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 20 | 64
  Male | 10 | 9 | 11 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 4
  Not Hispanic or Latino | 31 | 28 | 31 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 6 | 10 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 2 | 7
  White | 22 | 20 | 19 | 61
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Severity of Alopecia Tool Score at Week 24 in Placebo-Controlled Treatment Period
Description: The Severity of Alopecia Tool (SALT) score is a quantitative rating scale for measuring the severity of alopecia areata based on the amount of terminal hair loss in each of the 4 quadrants of the scalp: back region, top region, left and right regions of the scalp. To calculate a SALT score, the degree of scalp hair loss, as a percentage of each scalp region affected, is determined. Each region is multiplied by it's respective weighting factor (percentage surface area of the scalp in that area; back region [24%], top region [40%], left region [18%] and, right region [18%]), in order to achieve a subtotal for each region. The SALT score is the sum of the scalp hair loss in each area (sum of the subtotals). The score ranges from 0 to 100, the higher score reflects high severity of alopecia areata.
Time Frame: Baseline (Day 1) and Week 24
Population: Randomized population includes all participants who were in the enrolled population (who signed informed consent form) and were randomized using Interactive Response Technology (IRT).
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Placebo-Controlled: Deucravacitinib 6 mg QD: Participants with alopecia areata received deucravacitinib 6 mg tablet orally once daily (QD) from Day 1 to Week 24 in Placebo-controlled Period.
- Placebo-Controlled: Deucravacitinib 6 mg BID: Participants with alopecia areata received deucravacitinib 6 mg tablet orally twice daily (BID) from Day 1 to Week 24 in Placebo-controlled Period.
Arm/Group | Placebo-Controlled: Deucravacitinib 6 mg QD | Placebo-Controlled: Deucravacitinib 6 mg BID | Placebo
Number analyzed (Participants) | 32 | 31 | 31
Score on a Scale | -5.809 (13.3892) | 1.027 (14.7258) | -7.302 (17.8732)

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events in Placebo-Controlled Period
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization. Adverse event of interest included herpes zoster, malignancy, opportunistic infection or tuberculosis infection.
Time Frame: From first dose (Day 1) and up to 30 days after last dose for all participants (up to approximately 28 weeks)
Population: Safety population included all participants who were in the randomized population and received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled: Deucravacitinib 6 mg QD | Placebo-Controlled: Deucravacitinib 6 mg BID | Placebo
Number analyzed (Participants) | 32 | 31 | 31
Participants
  Treatment Emergent Adverse Events | 25 | 28 | 20
  Serious Treatment Emergent Adverse Events | 1 | 1 | 0
  Treatment Emergent Adverse Events Leading to Discontinuation of Study | 1 | 3 | 0
  TEAE of Interest-Herpes Zoster | 1 | 0 | 0
  TEAE of Interest-Malignancy-Bowen's Disease) | 0 | 1 | 0
  TEAE of Interest-Malignancy-Nodular lymphocyte predominant Hodgkin Lymphoma | 0 | 1 | 0
  TEAE of Interest - Opportunistic Infections | 0 | 0 | 0
  TEAE of Interest - Tuberculosis Infection | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events in Active Treatment Period
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization. Adverse event of interest included Herpes zoster, malignancy, opportunities infection or tuberculosis infection.
Time Frame: From first dose (Day 1) of Week 25 and up to 30 days after last dose for all participants (up to approximately 28 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Active Treatment Period: Deucravacitinib 6 mg QD: Participants initially randomized to deucravacitinib 6 mg QD in placebo-controlled period continued on their assigned dosage in Active Treatment Period till Week 52.
- Active Treatment Period: Deucravacitinib 6 mg BID: Participants initially randomized to deucravacitinib 6 mg BID in Placebo-controlled Period continued on their assigned dosage in Active Treatment Period till Week 52.
- Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg BID: Participants initially randomized to receive placebo in Placebo-controlled period were re-randomized to this arm at the Week 24 visit. Participants in this arm received 6 mg deucravacitinib tablet orally BID till Week 52 in Active Treatment Period.
Arm/Group | Active Treatment Period: Deucravacitinib 6 mg QD | Active Treatment Period: Deucravacitinib 6 mg BID | Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD | Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg BID
Number analyzed (Participants) | 32 | 26 | 16 | 15
Participants
  Treatment Emergent Adverse Events | 21 | 17 | 13 | 14
  Serious Treatment Emergent Adverse Events | 0 | 1 | 0 | 0
  Treatment Emergent Adverse Events Leading to Discontinuation of Study | 1 | 0 | 1 | 0
  TEAE of Interest-Herpes Zoster | 0 | 0 | 0 | 0
  TEAE of Interest-Malignancy-Bowen's Disease | 0 | 0 | 0 | 0
  TEAE of Interest-Malignancy-Nodular lymphocyte predominant Hodgkin Lymphoma | 0 | 0 | 0 | 0
  TEAE of Interest - Opportunistic Infections | 0 | 0 | 0 | 0
  TEAE of Interest - Tuberculosis Infection | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Worst Toxicity Grade Change From Baseline to Grade 3/Grade 4 in Laboratory Test Results as Per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 in Placebo-Controlled Period
Description: Blood samples were collected for assessment of laboratory test results. All abnormalities were graded as per CTCAE v5.0 on a scale from 1 to 4, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization.
Time Frame: From first dose (Day 1) through Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled: Deucravacitinib 6 mg QD | Placebo-Controlled: Deucravacitinib 6 mg BID | Placebo
Number analyzed (Participants) | 32 | 31 | 31
Participants
  HEMOGLOBIN, LOW | 0 | 0 | 0
  PLATELET COUNT, LOW | 0 | 0 | 0
  LEUKOCYTES, LOW | 0 | 0 | 0
  ALANINE AMINOTRANSFERASE (ALT), HIGH | 0 | 0 | 0
  ALKALINE PHOSPHATASE (ALP), HIGH | 0 | 0 | 0
  ASPARTATE AMINOTRANSFERASE (AST), HIGH | 0 | 0 | 0
  BILIRUBIN, TOTAL, HIGH | 0 | 0 | 0
  CREATININE, ENZYMATIC, HIGH | 0 | 0 | 0
  ALBUMIN, LOW | 0 | 0 | 0
  CALCIUM, LOW | 0 | 0 | 0
  CALCIUM, HIGH | 0 | 0 | 0
  CHOLESTEROL, TOTAL (TC), HIGH | 0 | 0 | 0
  CREATINE KINASE (CK), HIGH | 0 | 1 | 2
  GLUCOSE, LOW | 0 | 0 | 0
  POTASSIUM, LOW | 0 | 0 | 0
  POTASSIUM, HIGH | 0 | 0 | 0
  SODIUM, LOW | 0 | 0 | 0
  SODIUM, HIGH | 0 | 0 | 0
  TRIGLYCERIDES, HIGH | 0 | 0 | 0
  GLUCOSE FASTING, LOW | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Worst Toxicity Grade Change From Baseline to Grade 3/Grade 4 in Laboratory Test Results as Per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 in in Active Treatment Period
Description: Blood samples were collected for assessment of laboratory test results. All abnormalities are graded as per CTCAE v5.0 on a scale from 1 to 4, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization.
Time Frame: From Week 25 to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Period: Deucravacitinib 6 mg QD | Active Treatment Period: Deucravacitinib 6 mg BID | Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD | Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg BID
Number analyzed (Participants) | 32 | 26 | 16 | 15
Participants
  HEMOGLOBIN, LOW | 0 | 0 | 0 | 0
  PLATELET COUNT, LOW | 0 | 0 | 0 | 0
  LEUKOCYTES, LOW | 0 | 0 | 0 | 0
  ALANINE AMINOTRANSFERASE (ALT), HIGH | 0 | 0 | 0 | 0
  ALKALINE PHOSPHATASE (ALP), HIGH | 0 | 0 | 0 | 0
  ASPARTATE AMINOTRANSFERASE (AST), HIGH | 0 | 0 | 0 | 0
  BILIRUBIN, TOTAL, HIGH | 0 | 0 | 0 | 0
  CREATININE, ENZYMATIC, HIGH | 0 | 0 | 0 | 0
  ALBUMIN, LOW | 0 | 0 | 0 | 0
  CALCIUM, LOW | 0 | 0 | 0 | 0
  CALCIUM, HIGH | 0 | 0 | 0 | 0
  CHOLESTEROL, TOTAL (TC), HIGH | 0 | 0 | 0 | 0
  CREATINE KINASE (CK), HIGH | 0 | 0 | 0 | 0
  GLUCOSE, LOW | 0 | 0 | 0 | 0
  POTASSIUM, LOW | 0 | 0 | 0 | 0
  POTASSIUM, HIGH | 0 | 0 | 0 | 0
  SODIUM, LOW | 0 | 0 | 0 | 0
  SODIUM, HIGH | 0 | 0 | 0 | 0
  TRIGLYCERIDES, HIGH | 0 | 0 | 0 | 0
  GLUCOSE FASTING, LOW | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Marked Electrocardiogram Abnormalities in Placebo-Controlled Period
Description: A 12-lead ECG was performed after the participant remained supine for at least 5 minutes prior to the ECG. The ECG results read by the principal study investigator or a qualified and delegated designee as per local requirements
Time Frame: First dose (Day 1) to Week 24
Population: Safety population included all participants who were in the randomized population and received at least 1 dose of study intervention. Participants with ECG measurements at specified timepoints are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled: Deucravacitinib 6 mg QD | Placebo-Controlled: Deucravacitinib 6 mg BID | Placebo
Number analyzed (Participants) | 32 | 29 | 31
Participants
  QTCF 450 -< 480 MILLISECONDS (MSEC) | 0 | 2 | 1
  QTCF 480 -< 500 MSEC | 0 | 0 | 0
  QTCF >= 500 MSEC | 0 | 0 | 0
  QTCF 30 < CHANGE FROM BASELINE <= 60 MSEC | 0 | 1 | 0
  QTCF CHANGE FROM BASELINE > 60 MSEC | 0 | 0 | 0
  PR INTERVAL >= 200 MSEC | 2 | 0 | 1
  QRS INTERVAL >= 120 MSEC | 0 | 0 | 1

7. Primary Outcome: Number of Participants With Marked Electrocardiogram Abnormalities in Active Treatment Period
Description: A 12-lead ECG should be performed after the participant has remained supine for at least 5 minutes prior to the ECG. The ECG results will be read by the principal study investigator or a qualified and delegated designee as per local requirements
Time Frame: Week 25 to Week 52
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Period: Deucravacitinib 6 mg QD | Active Treatment Period: Deucravacitinib 6 mg BID | Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD | Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg BID
Number analyzed (Participants) | 28 | 19 | 14 | 14
Participants
  QTCF 450 -< 480 MILLISECONDS (MSEC) | 0 | 0 | 0 | 0
  QTCF 480 -< 500 MSEC | 0 | 0 | 0 | 0
  QTCF >= 500 MSEC | 0 | 0 | 0 | 0
  QTCF 30 < CHANGE FROM BASELINE <= 60 MSEC | 1 | 1 | 1 | 1
  QTCF CHANGE FROM BASELINE > 60 MSEC | 0 | 0 | 0 | 0
  PR INTERVAL >= 200 MSEC | 1 | 0 | 1 | 1
  QRS INTERVAL >= 120 MSEC | 1 | 0 | 1 | 0

8. Primary Outcome: Number of Participants With Abnormalities in Marked Vital Signs in Placebo-Controlled Period
Description: Vital signs such as systolic blood pressures (SBP), diastolic blood pressure (DBP) and heart rate were assessed. The evaluation of the marked abnormality criteria is based on participants highest change from baseline in the period. Blood pressure and heart rate were to be measured after the participant has been resting quietly for at least 5 minutes.
Time Frame: First dose (Day 1) to Week 24
Population: Safety population included all participants who were in the randomized population and received at least 1 dose of study intervention. Participants with vital sign measurements at specified timepoints are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled: Deucravacitinib 6 mg QD | Placebo-Controlled: Deucravacitinib 6 mg BID | Placebo
Number analyzed (Participants) | 32 | 30 | 31
Participants
  HEART RATE > 100 BPM AND CHANGE FROM BASELINE > 30 BPM | 0 | 1 | 0
  HEART RATE < 55 BPM AND CHANGE FROM BASELINE < -15 BPM | 1 | 0 | 0
  SBP >140 MM HG AND CHANGE FROM BASELINE > 20 MM HG | 1 | 4 | 1
  SBP <90 MM HG AND CHANGE FROM BASELINE < -20 MM HG | 0 | 0 | 1
  DBP >90 MM HG AND CHANGE FROM BASELINE > 10 MM HG | 3 | 0 | 1
  DBP <55 MM HG AND CHANGE FROM BASELINE < -10 MM HG | 0 | 0 | 1

9. Primary Outcome: Number of Participants With Abnormalities in Marked Vital Signs in Active Treatment Period
Description: Vital signs such as systolic blood pressures (SBP), diastolic blood pressure (DBP) and heart rate were assessed. The evaluation of the marked abnormality criteria is based on participants highest change from baseline in the period. Blood pressure and heart rate were to be measured after the participant had been resting quietly for at least 5 minutes.
Time Frame: Week 25 to Week 52
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Period: Deucravacitinib 6 mg QD | Active Treatment Period: Deucravacitinib 6 mg BID | Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD | Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg BID
Number analyzed (Participants) | 32 | 26 | 16 | 15
Participants
  HEART RATE > 100 BPM AND CHANGE FROM BASELINE > 30 BPM | 0 | 0 | 0 | 1
  HEART RATE < 55 BPM AND CHANGE FROM BASELINE < -15 BPM | 1 | 1 | 0 | 0
  SBP >140 MM HG AND CHANGE FROM BASELINE > 20 MM HG | 1 | 1 | 0 | 1
  SBP <90 MM HG AND CHANGE FROM BASELINE < -20 MM HG | 0 | 0 | 0 | 0
  DBP >90 MM HG AND CHANGE FROM BASELINE > 10 MM HG | 0 | 1 | 0 | 3
  DBP <55 MM HG AND CHANGE FROM BASELINE < -10 MM HG | 1 | 0 | 1 | 0

10. Secondary Outcome: Percentage of Participants Achieving a ≥ 50% Reduction in Severity of Alopecia Tool (SALT) Score (SALT50 Response) From Baseline at Week 24
Description: The Severity of Alopecia Tool (SALT) score is a quantitative rating scale for measuring the severity of alopecia areata based on the amount of terminal hair loss in each of the 4 quadrants of the scalp; back region, top region, left and right regions of the scalp. To calculate a SALT score, the degree of scalp hair loss, as a percentage of each scalp region affected, is determined. Each region is multiplied by its respective weighting factor (percentage surface area of the scalp in that area; Back region [24%], Left Region [18%], Right Region [18%], Top Region [40%]), in order to achieve a subtotal for each region. The SALT score is the sum of the scalp hair loss in each area (sum of the subtotals). The score ranges from 0 to 100, the higher score reflects high severity of alopecia areata. SALT50 response indicates at least a 50% improvement from baseline in the SALT score at a particular time point, indicating 50% hair regrowth.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo-Controlled: Deucravacitinib 6 mg QD | Placebo-Controlled: Deucravacitinib 6 mg BID | Placebo
Number analyzed (Participants) | 32 | 31 | 31
Percentage of participants | 3.1 | 0 | 6.5

11. Secondary Outcome: Percentage of Participants Achieving a Severity of Alopecia Tool (SALT) Score ≤20 at Week 24
Description: The Severity of Alopecia Tool (SALT) score is a quantitative rating scale for measuring the severity of alopecia areata based on the amount of terminal hair loss in each of the 4 quadrants of the scalp; back region, top region, left and right regions of the scalp. To calculate a SALT score, the degree of scalp hair loss, as a percentage of each scalp region affected, is determined. Each region is multiplied by its respective weighting factor (percentage surface area of the scalp in that area; Back region [24%], Left Region [18%], Right Region [18%], Top Region [40%]), in order to achieve a subtotal for each region. The SALT score is the sum of the scalp hair loss in each area (sum of the subtotals). The score ranges from 0 to 100, the higher score reflects high severity of alopecia areata. percentage of participants achieving an absolute SALT score ≤ 20, indicates ≤ 20% scalp hair loss.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo-Controlled: Deucravacitinib 6 mg QD | Placebo-Controlled: Deucravacitinib 6 mg BID | Placebo
Number analyzed (Participants) | 32 | 31 | 31
Percentage of participants | 3.1 | 0 | 0

12. Secondary Outcome: Percentage of Participants Achieving an Alopecia Areata Investigator Global Assessment (AA-IGA) Score of 0 or 1 at Week 24 With at Least a 2-Point Change From Baseline
Description: The AA-IGA utilizes a 5-points scale, in which the investigator assesses scalp hair loss based on the SALT assessment. The AA-IGA measures alopecia areata severity at a single point in time(without taking into account the baseline disease condition).The participant's scalp hair loss, as it look at the time of evaluation is scored as none (0) (0% scalp hair loss), limited (1) (1%-20% scalp hair loss), moderate (2) (21%-49% scalp hair loss), severe (3) (50%-94% scalp hair loss), or very severe (4)(95%-100 % scalp hair loss).
Time Frame: Baseline (Day 1) and week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo-Controlled: Deucravacitinib 6 mg QD | Placebo-Controlled: Deucravacitinib 6 mg BID | Placebo
Number analyzed (Participants) | 32 | 31 | 31
Percentage of participants | 3.1 | 0 | 0

13. Primary Outcome: Number of Participants With Abnormalities in Targeted Physical Examination Parameters in Placebo-Controlled Period
Description: Participants were assessed for abnormalities in targeted physical parameters.
Time Frame: First dose (Day 1) to Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled: Deucravacitinib 6 mg QD | Placebo-Controlled: Deucravacitinib 6 mg BID | Placebo
Number analyzed (Participants) | 32 | 31 | 31
Participants
  Abdomen | 0 | 0 | 1
  Extremities | 0 | 1 | 1
  General Appearance | 1 | 1 | 0
  Genitourinary | 1 | 0 | 0
  Head, Eyes, Ears, Nose, Throat | 3 | 6 | 2
  Lymph Nodes | 0 | 0 | 0
  Mouth | 3 | 0 | 0
  Musculoskeletal | 1 | 1 | 0
  Neck | 0 | 0 | 0
  Neurological | 2 | 0 | 1
  Psychiatric | 1 | 0 | 1
  Respiratory | 0 | 1 | 1
  Skin | 9 | 14 | 6
  Other | 1 | 1 | 0

14. Primary Outcome: Number of Participants With Abnormalities in Targeted Physical Examination Parameters in Active Treatment Parameters
Description: Participants were assessed for abnormalities in targeted physical parameters.
Time Frame: Week 25 to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Active Treatment Period: Placebo Followed bDeucravacitinib 6 mg BID: Participants initially randomized to receive placebo in Placebo-controlled Period were re-randomized to this arm at the Week 24 visit. Participants in this arm received 6 mg deucravacitinib tablet orally BID till Week 52 in Active Treatment Period.
Arm/Group | Active Treatment Period: Deucravacitinib 6 mg QD | Active Treatment Period: Deucravacitinib 6 mg BID | Active Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD | Active Treatment Period: Placebo Followed bDeucravacitinib 6 mg BID
Number analyzed (Participants) | 32 | 26 | 16 | 15
Participants
  Abdomen | 0 | 3 | 0 | 0
  Extremities | 0 | 1 | 0 | 0
  General Appearance | 0 | 0 | 0 | 0
  Genitourinary | 1 | 1 | 0 | 0
  Head, Eyes, Ears, Nose, Throat | 0 | 5 | 2 | 2
  Lymph Nodes | 0 | 1 | 0 | 0
  Mouth | 2 | 1 | 1 | 2
  Musculoskeletal | 1 | 2 | 1 | 0
  Neck | 0 | 1 | 0 | 0
  Neurological | 0 | 0 | 0 | 0
  Other | 2 | 2 | 0 | 4
  Psychiatric | 0 | 0 | 0 | 1
  Respiratory | 1 | 3 | 0 | 2
  Skin | 8 | 6 | 5 | 8

ADVERSE EVENTS:
Time Frame: All cause mortality was collected from Week 0 to Week 52. Serious AEs were collected from informed consent form signing (Week -4) and up to 30 days after last dose for all participants (up to approximately 32 weeks and 28 weeks in Placebo-controlled and Active Treatment Period respectively). Non Serious AEs were collected from first dose (Day 1) and up to 30 days after last dose (up to approximately 28 weeks for each Placebo-controlled and Active Treatment Period).
Description: Safety population included all participants who were in the randomized population and received at least 1 dose of study intervention.
Groups:
- Active-Treatment Period: Deucravacitinib 6 mg QD: Participants initially randomized to deucravacitinib 6 mg QD in Placebo-controlled Period continued on their assigned dosage in Active Treatment Period till Week 52.
- Active-Treatment Period: Deucravacitinib 6 mg BID: Participants initially randomized to deucravacitinib 6 mg BID in Placebo-controlled Period continued on their assigned dosage in Active Treatment Period till Week 52.
- Active-Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD: Participants initially randomized to receive placebo in Placebo-controlled Period were re-randomized to this arm at the Week 24 visit. Participants in this arm received 6 mg deucravacitinib QD tablet orally till Week 52 in Active Treatment Period.
Arm/Group | Placebo-Controlled: Deucravacitinib 6 mg QD | Placebo-Controlled: Deucravacitinib 6 mg BID | Placebo | Active-Treatment Period: Deucravacitinib 6 mg QD | Active-Treatment Period: Deucravacitinib 6 mg BID | Active-Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD | Active-Treatment Period: Placebo Followed by Deucravacitinib 6 mg BID
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31 | 0/31 | 0/32 | 0/26 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/32 | 1/31 | 0/31 | 0/32 | 1/26 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 24/32 | 26/31 | 16/31 | 15/32 | 14/26 | 13/16 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled: Deucravacitinib 6 mg QD (N=32) | Placebo-Controlled: Deucravacitinib 6 mg BID (N=31) | Placebo (N=31) | Active-Treatment Period: Deucravacitinib 6 mg QD (N=32) | Active-Treatment Period: Deucravacitinib 6 mg BID (N=26) | Active-Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD (N=16) | Active-Treatment Period: Placebo Followed by Deucravacitinib 6 mg BID (N=15)
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nodular lymphocyte predominant Hodgkin Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled: Deucravacitinib 6 mg QD (N=32) | Placebo-Controlled: Deucravacitinib 6 mg BID (N=31) | Placebo (N=31) | Active-Treatment Period: Deucravacitinib 6 mg QD (N=32) | Active-Treatment Period: Deucravacitinib 6 mg BID (N=26) | Active-Treatment Period: Placebo Followed by Deucravacitinib 6 mg QD (N=16) | Active-Treatment Period: Placebo Followed by Deucravacitinib 6 mg BID (N=15)
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1
Amalgam tattoo (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 3 | 4 | 1 | 0 | 2 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 3 | 1 | 0 | 1 | 1 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 2 | 0 | 2 | 2 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 5 | 6 | 1 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 1 | 2 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 8 | 0 | 2 | 6 | 2 | 1
Oral herpes (Infections and infestations) | 1 | 2 | 2 | 0 | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 0 | 2 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 4 | 4 | 5 | 4 | 4
Urinary tract infection (Infections and infestations) | 1 | 3 | 0 | 2 | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 1 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 3 | 3 | 3 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 5 | 4 | 3 | 0 | 0 | 3 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT05556265/Prot_SAP_000.pdf